CLINICAL TRIAL: NCT03288935
Title: Trauma Informed Care for Refugee Newcomers in Virginia: A Factorial Design of Effectiveness-Implementation Hybrid Research
Brief Title: Trauma Informed Care for Newly Resettled Refugees
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A substantial decrease in refugee arrivals in Virginia didn't allow the investigator to continue the study as planned.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: HM20011389
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mental Stress; Emotional Stress
Keywords: refugee; trauma-informed case management (TICM); trauma-informed cultural orientation (TICO); PTSD; depression; refugee resettlement
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (TICM only) (Active Comparator): Assigned to TICM group after reception & placement.
  Interventions: Behavioral: TICM
- Group 2 (TICO only) (Active Comparator): Assigned to TICO group after reception & placement.
  Interventions: Behavioral: TICO
- Group 3 (TICM & TICO) (Active Comparator): Assigned to both TICM and TICO group after reception & placement.
  Interventions: Behavioral: TICM; Behavioral: TICO
- Group 4 (None) (No Intervention): No additional intervention after reception & placement

INTERVENTIONS:
Behavioral: TICM — The TICM will be designed to include the seven domains of trauma-informed care articulated by SAMHSA (2014): 1) early screening and comprehensive assessment; 2) consumer driven care and services; 3) trauma-informed, responsive and educated workforce; 4) emerging and evidence-informed best practices; 5) safe and secure environments; 6) trauma-informed community partnerships; and 7) a performance monitoring system. The trained agency case managers and staff will provide the TICM to 50 newly resettled refugees during their regular R&P service period (i.e., 60 days).
  Arms: Group 1 (TICM only); Group 3 (TICM & TICO)
Behavioral: TICO — The community-based TICO will be based on the Im's CHW that comprises 8 sessions (2 hour per session), co-facilitated by trained refugee peer mentors and community service providers. The TICO sessions will include interactive sessions on healthy eating, healthy body and healthy mind, acculturation & resettlement stress, understanding trauma and stress, healthy coping, helping others, and community building.
  Arms: Group 2 (TICO only); Group 3 (TICM & TICO)

SUMMARY:
The main purpose of this study is to evaluate early-phase interventions for refugee wellness promotion and build evidence for dissemination of the intervention model and curricula through refugee resettlement programs, local and national.

DETAILED DESCRIPTION:
This study will examine the main effects of trauma-informed case management (TICM) and trauma-informed cultural orientation (TICO) interventions, respectively, in reducing resettlement distress and increasing coping capacity, which will improve emotional wellness and social adaptation and thus resettlement outcomes. This project will also test the interaction effects of two-tiered intervention model, discerning effective and ineffective components of the intervention model. Differences in effects across intervention conditions may inform how improvement in what outcomes or which phase can affect refugees' wellness and adjustment over time.

ELIGIBILITY:
Inclusion Criteria:

* Refugee adults who arrive in Richmond or Charlottesville between January and February 2018

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Change in resettlement distress | Baseline to 6 months
  Penn State Worry Questionnaire, which captures pervasiveness, excessiveness, and uncontrollability of worry. Scores range from 16 to 80 with higher values indicating more worry.

SECONDARY OUTCOMES:
Change in emotional well-being | Baseline to 6 months
  Refugee Health Screener-15, a 75 item screening tool with lower scores indicating better well-being
Resettlement Outcomes | Baseline to 6 months
  Post-Migration Living Difficulties, a self-assessment tool which measures adverse post -migration experiences in five different domains, included two related asylum-seeking factors. Scores range from 23 to 115 with higher values indicating more serious problems.
Change in Social Adaptation | Baseline to 6 months
  Social Adaptation Self-evaluation Scale. Scores range from 0 to 63 with higher values indicating better social adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Hyojin Im, PhD, Principal Investigator — Virginia Commonwealth Univeristy
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States